CLINICAL TRIAL: NCT05503862
Title: Randomized Controlled Trial of Home Semen Testing in Men Beginning Attempts to Conceive
Brief Title: Home Semen Testing in Men Beginning Attempts to Conceive
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Joshua Halpern, Assistant Professor, Department of Urology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00216874
Record Dates: First submitted 2022-07-12; First posted 2022-08-17 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized to one of two arms: standard of care office-based pathway or the at home semen testing pathway utilizing the FDA, commercially approved YoSperm® device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm A (Experimental): At home semen testing via the YoSperm device
  Interventions: Device: YoSperm
- Arm B (No Intervention): Standard of Care

INTERVENTIONS:
Device: YoSperm — The purpose of the app is for at-home semen analysis including sperm motility concentration and sperm quality (YO Score) and compares the results to laboratory standards. We will be utilizing the YoSperm® technology in order for patients to send their semen analysis results directly from their device to their provider via secure email.
  Arms: Arm A

SUMMARY:
The overall objective of the proposed study is to enhance early detection of male factor infertility and reduce cost and morbidity associated with delayed diagnosis through development of a universal screening model based on home semen testing. The advent of inexpensive and accurate home semen testing has enabled a potential paradigm shift in the approach to male fertility evaluation. The investigator's central hypothesis is that universal home semen testing prior to attempts to conceive is easy for participants and can lead to reduced fertility-related anxiety and early detection of male factor infertility, thereby expediting evaluation and treatment for the couple while minimizing unnecessary cost and morbidity.

This study is specifically designed to assess the feasibility and utility of home semen testing for couples who are beginning attempts to conceive. First, the investigator will assess participants' ability to complete the home semen testing, ease of use, and obstacles encountered in doing so. Second, the investigator will examine the impact of home semen testing in fertility-related quality of life among couples beginning attempts to conceive, as well as ability of home semen testing to increase the diagnosis and treatment of male infertility in these couples.

ELIGIBILITY:
Inclusion Criteria:

* Natal males over the age of 18 with no prior children who are interested in future fertility
* Current female partner
* Not attempting to conceive for more than 3 months
* Willing to sign the Informed Consent Form
* Able to read, understand, and complete patient questionnaires, pain texts, and medication diary.
* Ownership or accessibility of a smart phone or electronic device that is compatible with the YoSperm® device

Exclusion Criteria

* Prior semen testing
* History of male infertility, Klinefelter syndrome, undescended testis, or chemotherapy
* Female partner with history of infertility
* Female partner with irregular menstrual periods

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Was the home semen testing completed- yes/no? | At Day 0 post randomization
  To assess if participants randomized to the home semen testing utilize the YoSperm device to complete the home semen testing.
Change in fertility-related World Health organization-5 Well-Being Index (WHO-5). | 12 months
  To assess participant well-being over the course of the study.
Subsequent pursuit of formal male infertility evaluation via the follow-up Fertility Questionnaire. | 12 months
  To evaluate the participant's fertility over the course of the study.
Change in fertility-related Fertility Quality of Life Questionnaire (FertiQoL) | 12 months
  To assess participant's fertility quality of life over the course of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Department of Urology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT05503862/Prot_000.pdf
  • Informed Consent Form (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/62/NCT05503862/ICF_001.pdf